CLINICAL TRIAL: NCT01000350
Title: Intravenous Saline on Exercise Tolerance in Orthostatic Intolerance
Brief Title: Intravenous (IV) Saline and Exercise in Postural Tachycardia Syndrome (POTS)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Satish R. Raj, Adjunct Associate Professor of Medicine, Vanderbilt University Medical Center
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 090942
Record Dates: First submitted 2009-10-21; First posted 2009-10-23 (Estimated); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Postural Tachycardia Syndrome
Keywords: orthostatic intolerance; exercise capacity; tachycardia; POTS
MeSH Terms: conditions — Postural Orthostatic Tachycardia Syndrome; Orthostatic Intolerance; Tachycardia | interventions — Sodium Chloride; Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise Post Saline (Experimental): Saline infusion 1L hours before exercise test
  Interventions: Drug: Saline
- Placebo (Placebo Comparator): Placebo given prior to exercise test
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Saline — IV Normal Saline infused over 30-60 minutes given 3-6 hours PRIOR to exercise study
  Other Names: Normal Saline; 0.9% saline
  Arms: Exercise Post Saline
Other: Placebo — Placebo x1 lactose tablet
  Arms: Placebo

SUMMARY:
The investigators will test whether an intravenous infusion of saline (salt water) will improve the exercise capacity in patients with postural tachycardia syndrome (POTS).

ELIGIBILITY:
Inclusion Criteria:

* Meet diagnostic criteria of Postural Tachycardia Syndrome (POTS) 28
* Age between 18-65 years
* Male and female are eligible (although the majority of POTS patients are female).
* Able and willing to provide informed consent

Exclusion Criteria:

* Presence of medical conditions that can explain postural tachycardia (e.g., acute dehydration, medications)
* Pregnancy
* Other factors which in the investigator's opinion would prevent the subject from completing the protocol.
* Patients who are bedridden or chair-ridden

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2009-10; Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Difference in VO2max between saline day and placebo day | Within 2 week
  VO2max will be measured hours after saline and after placebo. The 2 interventions will be less than 2 weeks apart.

SECONDARY OUTCOMES:
Exercise capacity/Maximal Load (Watts) during peak VO2 | Less than 2 weeks
  Maximal exercise load will be measured hours after saline and after placebo. The 2 interventions will be less than 2 weeks apart.
Cardiac output between exercise tests (inert gas rebreathing technique) | 2-10 Days between exercise tests

CONTACTS AND LOCATIONS:
Overall Officials: Satish R Raj, MD MSCI, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States

REFERENCES:
- [Background] Raj SR, Biaggioni I, Yamhure PC, Black BK, Paranjape SY, Byrne DW, Robertson D. Renin-aldosterone paradox and perturbed blood volume regulation underlying postural tachycardia syndrome. Circulation. 2005 Apr 5;111(13):1574-82. doi: 10.1161/01.CIR.0000160356.97313.5D. Epub 2005 Mar 21. PMID 15781744